CLINICAL TRIAL: NCT00697294
Title: Vitamin D Status and Impact on Bone Mineralization in Human Milk Fed Hispanic and Caucasian Infants
Brief Title: Impact of Vitamin D Status on Bones in Breastfed Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Steve Abrams, MD, Professor, Baylor College of Medicine
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: H-22293
Record Dates: First submitted 2008-06-03; First posted 2008-06-13 (Estimated); Last update posted 2011-12-05 (Estimated); Status verified 2011-12

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D deficiency; Infants; Breast feeding
MeSH Terms: conditions — Vitamin D Deficiency; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supplement (Experimental): Subjects will serve as their own control in this single-arm protocol. All subjects will receive 400 IU/day of vitamin D as the intervention. Comparisons will be made between Caucasian and Hispanic infants.
  Interventions: Dietary Supplement: Tri-Vi-Sol

INTERVENTIONS:
Dietary Supplement: Tri-Vi-Sol — All subjects will begin vitamin D supplementation at the first outpatient visit (at 1 week of life) and will continue through the second outpatient visit (at 3 months of age). Dosage will be 400 IU/day of vitamin D in the form of Tri-Vi-Sol vitamin drops.
  Other Names: ADC drops

SUMMARY:
Vitamin D deficiency is widespread and linked to decreased bone mineral content. Little data exists regarding the vitamin D status and the relationship of 25-hydroxyvitamin D (25-OHD) status to functional bone health outcomes in Hispanic infants. To evaluate this, we plan an observational cohort of full term, healthy, exclusively breastfed Hispanic and Caucasian infants. We hypothesize serum 25-OHD measured in cord blood will be significantly lower in Hispanic than Caucasian infants, with 25-OHD less than 20 ng/mL found in at least 50% of Hispanic neonates. Secondary aims evaluate the relationship between 25-OHD levels and bone mineral status at baseline and after 3 months of 400 IU/day supplemental vitamin D3. Whole body bone density scan (DXA) and bone ultrasound (SOS U/S) will be measured shortly after birth, then again after supplementation. Data from this study will provide information needed to design further randomized trials and interventions.

DETAILED DESCRIPTION:
In recent years, severe vitamin D deficiency has resurfaced as a major public health concern. Nutritional rickets is widespread, and a recent report on this disease in Texas showed Hispanic children are at increased risk. Long-term follow-up has demonstrated that vitamin D deficient infants are more likely to have decreased bone mineral status in late childhood. Additionally, vitamin D deficiency has been linked to changes in fetal "imprinting" and increased susceptibility to autoimmune diseases, immune deficiency, and malignancy. At birth, an infant's vitamin D status is entirely dependent on the vitamin D status of the mother. Many studies have shown vitamin D deficiency is very common in mother-child pairs, especially in dark-skinned individuals. However, few data exist regarding the vitamin D status in Hispanic infants. Low milk intakes and decreased sun exposure with urbanization makes this a very high-risk group among infants in Texas.

Potential subjects will be identified by study personnel in labor and delivery at St. Luke's and Ben Taub Hospitals and in the normal newborn nurseries. The parent/guardian will be approached and the study will be explained in full. A time for questions will be allowed. Once the parent/guardian agrees to his/her child's participation, an informed written consent form will be signed. Subject confidentiality will be maintained within limits of the law. All names and personal information will be accessed only by the investigators and authorized personnel. There will be no possibility of coercion as subjects will not have any relationship of dependency with the investigators.

A cohort of Hispanic and Caucasian infants will be recruited and followed. Other ethnic groups will not be excluded, but will not be analyzed in terms of the primary outcome. Race and ethnicity will be classified according to mother's self classification. The interventions will not differ between the groups.

This study includes 3 study visits:

1. Baseline inpatient visit at birth - while hospitalized to obtain consent, obtain cord blood sample, and mother to complete a questionnaire
2. 1 week after initial hospital discharge - first outpatient visit to obtain other baseline data (see below) and to start the vitamin D drops
3. At 3 mo of life - second outpatient visit to obtain final data (see below) and discontinue vitamin D drops

Visit 1 (Inpatient): After consent has been obtained and upon birth, cord blood will be obtained and analyzed using the Diasorin RIA for 25-OHD. In addition, serum ionized calcium and intact parathyroid hormone (PTH) concentration will be measured on cord blood. Mothers will be given a brief questionnaire to determine their risk of vitamin D deficiency (do they take vitamins, supplements, sun exposure). Follow-up outpatient appointments will be scheduled.

Visit 2 (First Outpatient Visit): Infants will have a speed of sound ultrasound (SOS U/S) and whole body dual-energy x-ray absorptiometry (DXA) performed at 1 week after hospital discharge. Supplements of 400 IU of vitamin D per day will be provided for all infants free of charge starting at the time of the body composition analysis (Vitamin D supplementation is recommended by the American Academy of Pediatrics for all infants who are exclusively breastfeeding).

Visit 3 (Second Outpatient Visit): Infants will return at three months of age and repeat measurements of serum 25-OHD, PTH, bone SOS U/S, and whole body DXA will be performed. At this time a second brief questionnaire will be given to the mother to assess the risks of vitamin D deficiency in the child. Vitamin D drops will be discontinued.

Between visits, investigators will call the family to check on breast feeding status.

At delivery, cord blood will be obtained and analyzed for 25-OHD, serum ionized calcium, and intact parathyroid hormone (PTH) concentration. At three months of age blood will be drawn for 25-OHD and PTH. The purpose of the blood draw is to assess the vitamin D status in the newborn infant. This is the primary aim of the study.

* 5 cc (one teaspoon) of cord blood will be obtained at visit 1, and 5 cc (one teaspoon) blood will be drawn from patient at the third visit (three months of age).
* Total = 2 teaspoons

There will be no study costs passed on the subject's family. Study investigations (laboratory, bone mineral assessment) will be paid for by the researchers. Costs for routine medical care, not associated with the study, but associated with delivery and hospitalization of the newly born child will be the responsibility of the family and their insurance company.

A total of 60 subjects will be enrolled in the protocol. Enrollment of 30 Hispanic infants and 30 Caucasian infants will provide a power > 80% to demonstrate a significantly lower cord 25-OHD concentration in Hispanic infants at p<0.05, the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Full term infants (37-42 weeks)
* Appropriate for gestational age
* Free of major congenital anomalies
* Born to mothers without a history of diabetes or chronic illness who intend to exclusively breastfeed

Exclusion Criteria:

* Any child who does not meet the above inclusion criteria
* Insufficient cord blood available to determine cord 25-hydroxyvitamin D status

Max Age: 2 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the relative frequency of vitamin D deficiency in human milk fed Hispanic compared to Caucasian newborn infants in Houston, Texas. | End of study

SECONDARY OUTCOMES:
To determine if infant vitamin D status is related to bone mineral status at birth | End of study
To determine the effects of vitamin D supplementation on 25-hydroxyvitamin D (25-OHD) concentration and bone mineral status vitamin D deficient and vitamin D replete infants at 3 months of age. | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Abrams, MD, Principal Investigator — Baylor College of Medicine
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - St Lukes Episcopal Hospital, Houston, Texas

REFERENCES:
- [Background] Shah M, Salhab N, Patterson D, Seikaly MG. Nutritional rickets still afflict children in north Texas. Tex Med. 2000 Jun;96(6):64-8. PMID 10876374
- [Background] Javaid MK, Crozier SR, Harvey NC, Gale CR, Dennison EM, Boucher BJ, Arden NK, Godfrey KM, Cooper C; Princess Anne Hospital Study Group. Maternal vitamin D status during pregnancy and childhood bone mass at age 9 years: a longitudinal study. Lancet. 2006 Jan 7;367(9504):36-43. doi: 10.1016/S0140-6736(06)67922-1. PMID 16399151
- [Background] McGrath J. Does 'imprinting' with low prenatal vitamin D contribute to the risk of various adult disorders? Med Hypotheses. 2001 Mar;56(3):367-71. doi: 10.1054/mehy.2000.1226. PMID 11359362
- [Background] Basile LA, Taylor SN, Wagner CL, Quinones L, Hollis BW. Neonatal vitamin D status at birth at latitude 32 degrees 72': evidence of deficiency. J Perinatol. 2007 Sep;27(9):568-71. doi: 10.1038/sj.jp.7211796. Epub 2007 Jul 12. PMID 17625571
- [Background] Dijkstra SH, van Beek A, Janssen JW, de Vleeschouwer LH, Huysman WA, van den Akker EL. High prevalence of vitamin D deficiency in newborn infants of high-risk mothers. Arch Dis Child. 2007 Sep;92(9):750-3. doi: 10.1136/adc.2006.105577. PMID 17715438
- [Background] Lee JM, Smith JR, Philipp BL, Chen TC, Mathieu J, Holick MF. Vitamin D deficiency in a healthy group of mothers and newborn infants. Clin Pediatr (Phila). 2007 Jan;46(1):42-4. doi: 10.1177/0009922806289311. PMID 17164508
- [Background] Brunvand L, Haga P, Tangsrud SE, Haug E. Congestive heart failure caused by vitamin D deficiency? Acta Paediatr. 1995 Jan;84(1):106-8. doi: 10.1111/j.1651-2227.1995.tb13499.x. PMID 7734890
- [Background] Brooke OG, Butters F, Wood C. Intrauterine vitamin D nutrition and postnatal growth in Asian infants. Br Med J (Clin Res Ed). 1981 Oct 17;283(6298):1024. doi: 10.1136/bmj.283.6298.1024. No abstract available. PMID 6794748
- [Background] Cockburn F, Belton NR, Purvis RJ, Giles MM, Brown JK, Turner TL, Wilkinson EM, Forfar JO, Barrie WJ, McKay GS, Pocock SJ. Maternal vitamin D intake and mineral metabolism in mothers and their newborn infants. Br Med J. 1980 Jul 5;281(6232):11-4. doi: 10.1136/bmj.281.6232.11. PMID 7407476
- [Background] Alfaham M, Woodhead S, Pask G, Davies D. Vitamin D deficiency: a concern in pregnant Asian women. Br J Nutr. 1995 Jun;73(6):881-7. doi: 10.1079/bjn19950093. PMID 7632669
- [Background] Datta S, Alfaham M, Davies DP, Dunstan F, Woodhead S, Evans J, Richards B. Vitamin D deficiency in pregnant women from a non-European ethnic minority population--an interventional study. BJOG. 2002 Aug;109(8):905-8. doi: 10.1111/j.1471-0528.2002.01171.x. PMID 12197370
- [Background] Waiters B, Godel JC, Basu TK. Perinatal vitamin D and calcium status of northern Canadian mothers and their newborn infants. J Am Coll Nutr. 1999 Apr;18(2):122-6. doi: 10.1080/07315724.1999.10718839. PMID 10204827
- [Background] Molla AM, Al Badawi M, Hammoud MS, Molla AM, Shukkur M, Thalib L, Eliwa MS. Vitamin D status of mothers and their neonates in Kuwait. Pediatr Int. 2005 Dec;47(6):649-52. doi: 10.1111/j.1442-200x.2005.02141.x. PMID 16354218
- [Background] Nicolaidou P, Hatzistamatiou Z, Papadopoulou A, Kaleyias J, Floropoulou E, Lagona E, Tsagris V, Costalos C, Antsaklis A. Low vitamin D status in mother-newborn pairs in Greece. Calcif Tissue Int. 2006 Jun;78(6):337-42. doi: 10.1007/s00223-006-0007-5. Epub 2006 Jul 7. PMID 16830197
- [Background] Abrams SA, Copeland KC, Gunn SK, Stuff JE, Clarke LL, Ellis KJ. Calcium absorption and kinetics are similar in 7- and 8-year-old Mexican-American and Caucasian girls despite hormonal differences. J Nutr. 1999 Mar;129(3):666-71. doi: 10.1093/jn/129.3.666. PMID 10082772
- [Background] Reasner CA 2nd, Dunn JF, Fetchick DA, Liel Y, Hollis BW, Epstein S, Shary J, Mundy GR, Bell NH. Alteration of vitamin D metabolism in Mexican-Americans. J Bone Miner Res. 1990 Jan;5(1):13-7. doi: 10.1002/jbmr.5650050105. PMID 2309575
- [Background] Looker AC, Orwoll ES, Johnston CC Jr, Lindsay RL, Wahner HW, Dunn WL, Calvo MS, Harris TB, Heyse SP. Prevalence of low femoral bone density in older U.S. adults from NHANES III. J Bone Miner Res. 1997 Nov;12(11):1761-8. doi: 10.1359/jbmr.1997.12.11.1761. PMID 9383679
- [Background] Zadshir A, Tareen N, Pan D, Norris K, Martins D. The prevalence of hypovitaminosis D among US adults: data from the NHANES III. Ethn Dis. 2005 Autumn;15(4 Suppl 5):S5-97-101. PMID 16315387
- [Background] Ashraf A, Mick G, Atchison J, Petrey B, Abdullatif H, McCormick K. Prevalence of hypovitaminosis D in early infantile hypocalcemia. J Pediatr Endocrinol Metab. 2006 Aug;19(8):1025-31. doi: 10.1515/jpem.2006.19.8.1025. PMID 16995588
- [Derived] Abrams SA, Hawthorne KM, Rogers SP, Hicks PD, Carpenter TO. Effects of ethnicity and vitamin D supplementation on vitamin D status and changes in bone mineral content in infants. BMC Pediatr. 2012 Jan 16;12:6. doi: 10.1186/1471-2431-12-6. PMID 22248486